CLINICAL TRIAL: NCT05668390
Title: A Multi-national Phase IIIb, Double-blind, Placebo-controlled Trial to Determine the Safety and Efficacy of STALORAL® Birch 300 IR in Children and Adolescents 5 to 17 yo With Birch Pollen-induced Allergic Rhinoconjunctivitis w/o Asthma
Brief Title: Safety and Efficacy of STALORAL® Birch 300 IR in a Paediatric Population With Birch Pollen-induced ARC w/o Asthma
Acronym: YOBI
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Stallergenes Greer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SL79.22
Record Dates: First submitted 2022-11-17; First posted 2022-12-29 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Allergic Rhinoconjunctivitis; Birch Pollen Allergy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STALORAL® Birch 300 IR (Experimental): 1. Escalation Phase:
     The escalation phase starts with 10 IR/mL solution the first 5 days (daily increase from 1 to 5 actuations) and switching to 300 IR/mL solution the next 5 days (daily increase from 1 to 5 actuations).
  2. Maintenance Phase:
  The maintenance phase takes place with 5 actuations of the active 300 IR/mL solution from Day 11 onwards
  Interventions: Drug: STALORAL® Birch 300 IR
- Placebo (Placebo Comparator): 1. Escalation Phase:
     The escalation phase starts with 10 IR/mL Placebo solution the first 5 days (daily increase from 1 to 5 actuations) and switching to 300 IR/mL Placebo solution the next 5 days (daily increase from 1 to 5 actuations).
  2. Maintenance Phase:
  The maintenance phase takes place with 5 actuations of the active 300 IR/mL Placebo solution from Day 11 onwards
  Interventions: Drug: STALORAL® Birch 300 IR

INTERVENTIONS:
Drug: STALORAL® Birch 300 IR — 2 treatment periods will consist of 2 steps: an escalation phase, where the treatment dose will gradually increase, followed by a maintenance phase.

SUMMARY:
Allergic rhinoconjunctivitis due to birch pollen is a seasonal problem which manifests as a combination of nasal symptoms (such as congestion, runny nose, sneezing, itching of the nose) and ocular symptoms (such as red, itchy and watery eyes). For several birch-allergic patients, allergic rhinoconjunctivitis occurs with an oral allergy syndrome.

The purpose of this study is to demonstrate the safety and efficacy of the study drug (STALORAL Birch 300 IR) in children and adolescents with birch pollen-induced allergic rhinoconjunctivitis, with or without asthma, when treated before and during the pollen season.

Approximately 699 children will participate in this study. The study will be conducted worldwide in approximately 80 medical sites in about 12 countries. The total duration of the study will be approximately 20 months.

DETAILED DESCRIPTION:
Birch pollen is a major cause of allergic rhinitis/allergic rhino-conjunctivitis in Europe and worldwide, with up to 100 million reported cases. Allergic rhinitis/allergic rhino-conjunctivitis (AR/ARC) is a chronic disorder of the upper airways that is caused by allergen exposure and the resulting inflammation of the nose and to a less extent, the eyes (allergic rhino-conjunctivitis). Rhinitis symptoms include sneezing, runny nose, nasal itching and nasal congestion and can be associated with conjunctivitis symptoms such as watery, red and/or itchy eyes. Current treatment are allergen avoidance, symptomatic pharmacotherapy, and Allergen Immunotherapy (AIT). However, avoidance measures are generally not effective. While symptomatic treatment can provide temporary relief from allergy symptoms, many patients remain uncontrolled.

The goal of this study is to demonstrate the clinical efficacy of an allergen immunotherapy (STALORAL Birch 300 IR) in children and adolescents from 5 to 17 years old with birch pollen-induced allergic rhinoconjunctivitis treated once daily pre- and co-seasonally over two consecutive birch pollen seasons on the average daily ARC Total Combined Score (TCS) during the season.

This study is a multi-national phase IIIb, double-blind, placebo-controlled study in which 699 participants will be enrolled in Europe for 20 months during two consecutive seasons.

Participants will begin STALORAL Birch 300 IR administration 3,5 months to 4,5 months prior to the birch pollen season (pre-seasonal treatment) and continue taking it for the duration of the season (co-seasonal treatment). There will approximately be 5 months of a treatment-free period prior to the next 3,5-month to 4-month pre-seasonal treatment period and co-seasonal treatment.

The analysis will be performed at the end of the Year 2.

ELIGIBILITY:
Inclusion Criteria:

1. Able to sign and date the informed consent/assent form prior to any trial-specific procedure. Patients may check a box on the assent form if they are unable to provide a signature.

   (Parents and/or authorised legal representative(s) will have to give written informed consent for minors in their custody)
2. Covered by a health insurance system as per local regulation.

   Demographics and Medical History
3. Aged ≥5 to ≤17 years old at the randomisation visit.
4. Documented, physician diagnosed, clinically relevant history of moderate to severe ARC induced by birch pollen (with or without asthma) despite having received treatment with symptom-relieving medication during at least 1 previous birch pollen season for ages 4 through 6 or at least 2 previous birch pollen seasons for ages 7 through 17 years at screening.
5. A Retrospective ARC Total Symptom Score (TSS) based on the previous birch pollen season at least 12 out of a maximum possible score of 18 AND a retrospective score of at least 30 on a general Visual Analog Scale (VAS) (0-100) on the severity of symptoms as evaluated by the patient or by the parent/authorised legal representative if the patient is not able to perform the assessment, at screening.

   Retrospective ARC TSS (0-18) is rated the same way as Daily Symptom Score (DSS) (0-18)

   Screening Tests and Evaluations
6. Positive Skin Prick Test (SPT) to Betula pendula at screening visit (the SPT is considered positive if it results in a wheal diameter ≥ 3.0 mm [with positive control (histamine) ≥ 3.0 mm and negative control = 0 mm]). The Sponsor will accept to include patients who have a documented positive SPT in their medical records if this SPT was performed during the previous 6 months preceding the screening visit at the same investigational site in which they are enrolled.
7. Positive specific Immunoglobulin E (IgE) to pollen allergens of Betula pendula at screening (CAP-RAST birch pollen allergens specific IgE ≥ 0.7 kU/L).
8. Negative urine pregnancy test on all female patients of childbearing potential or who have had their first menarche prior to randomisation.

   Lifestyle Considerations
9. Internet access at home or via a portable device so that patients or the parent/authorised legal representative can complete the e-Diary in a dedicated application on a mobile phone daily via internet. Patients will start scoring at randomisation, i.e., 4 months before the pollen season.

Exclusion Criteria:

Medical History

1. Any clinical deterioration of asthma (i.e., asthma exacerbation) that resulted in emergency procedure/treatment or treatment with systemic corticosteroids within 3 months prior to randomisation.
2. For patients ≥7 years old:

   Reduced lung function at randomisation defined as Forced Expiratory Volume in 1 second (FEV1) < 70% of the predicted value. For patients with asthma, this is assessed on the patient's usual asthma controller medication*. The following wash-out periods apply for as-needed asthma reliever medication: at least a 6-hour wash-out of Short-Acting Beta Agonists (SABAs), a 12-hour wash-out of Long-Acting Beta Agonists (LABAs),a 24-hour wash-out for ultra-LABAs and 5 days or 5 half-lives for inhaled corticosteroids.

   *In order to ensure that the asthmatic patients with a mild to moderate asthma status are controlled by treatment steps 1, 2 or 3 in accordance with the Global Initiative for Asthma (GINA 2022), the proper continuous asthma treatment i.e., "controller" is maintained. Only the asthma "reliever" medications must be stopped before performing spirometry. If an asthma medication is used as both "controller" and "reliever", such as inhaled corticosteroids (in combination with formoterol [LABA]), it must not be stopped before performing spirometry.

   Note: This criterion does not need to be fulfilled if the patient is <7 years old, as s/he cannot perform reproducible FEV1 manoeuvres despite coaching and is not considered as having a diagnosis of asthma.
3. Server or uncontrolled asthma with asthmatic therapies consistent with steps 4 or 5 as defined by Global Initiative for Asthma (GINA) 2022 received within 12 months prior to entry in the trial. Asthmatic patients with asthmatic therapies consistent with steps 1, 2 or 3 must be controlled (i.e. patients with controlled, mild and moderate asthma are eligible).
4. Severe oral inflammations such as oral lichen planus, oral ulcerations or oral mycosis.
5. Acute or chronic inflammatory or infectious upper airway diseases (excepted mild to moderate asthma) including recurrent acute or chronic sinusitis.

   Note: Patients with fever, flu or an upper respiratory tract infection at Visit 1 (screening visit) must be treated appropriately. They can be randomised at Visit 2 (randomisation visit) only if the infectious episode is resolved.
6. History of eosinophilic oesophagitis or with current severe or persistent gastroesophageal symptoms including dysphagia or chest pain that, in the opinion of the investigator, may constitute an increased safety concern.
7. A relevant history of systemic allergic reaction (e.g., anaphylaxis with cardiorespiratory symptoms, generalised urticaria or severe facial angioedema) that, in the opinion of the Investigator, may constitute an increased safety concern.
8. Any disease that prohibits the use of adrenaline (e.g., hyperthyroidism).
9. Any severe, uncontrolled disease that, upon Investigator judgment, could increase the risk for trial patients (including but not limited to cardiovascular insufficiency, any severe or unstable lung diseases, endocrine diseases, clinically significant renal or hepatic diseases, haematological disorders, diseases of the immune system including autoimmune diseases [upon the Investigator's judgment based on the benefit/risk assessment] and immune deficiencies of current clinical relevance, active malignancies).

   Screening Tests and Evaluations
10. A documented clinically relevant history of seasonal ARC symptoms caused by an allergen source, other than tree pollen from the birch homologous group, with a season overlapping the BPS.
11. A documented clinically relevant history of perennial ARC symptoms caused by an allergen source such as animal dander to which the patient is exposed during the BPS.
12. Any significant abnormal laboratory parameter or alteration in vital signs that could increase the risk for the patient, in the opinion of the Investigator.

    Medication
13. Ongoing treatment with prohibited treatment as listed in Section 8.2.3 or any allergen immunotherapy product including Specific Immunotherapy (SIT), or past full courses of SIT against birch pollen terminated for less than 5 years or past courses of SIT for other allergens terminated for less than 6 months prior to start of randomisation.
14. Patients requiring continuous treatment with systemic corticosteroids for any indications.
15. Patients requiring continuous treatment with β-blockers or with Monoamine Oxidase Inhibitors (MAOIs).
16. Treatment with an immunosuppressive (Anatomical Therapeutic Chemical code L04 or L01) within 3 months prior to the screening visit.
17. Hypersensitivity to any excipients of the IMP/placebo, or contraindication to the use of RMs (i.e., antihistamine and nasal corticosteroids).
18. Patients following a strict low sodium diet as the IMP treatment contains 590 mg of sodium chloride per vial in a 10 mL solution.
19. Inability to adhere to the washout periods as defined by the protocol, with respect to screening and to refrain from using the medications indicated until after the trial is complete.
20. Patients who would be likely to require prohibited concomitant therapy during the trial or who are anticipated to require using of such agents during the trial. Any medication given for an AE will be permitted.

Other

21. Breastfeeding females (lactating).

22. Sexually active females of childbearing potential or who have had their first menarche prior to randomisation who are not taking and/or willing to use either 1 highly effective contraceptive method or 2 clinically acceptable contraceptive methods until the end of the trial (depending on the local regulation):

* Acceptable highly effective methods of contraception

  1. Non-cyclic, stable dose (monophasic) combined oestrogen-progestin oral hormonal contraception associated with consistent inhibition of ovulation. Oral contraceptives containing oestrogens should be in stable use for at least 12 weeks prior to Screening.

  2. Desogestrel based progestin only contraception associated with consistent inhibition of ovulation; this includes oral, injectable, and implantable methods 3. Intravaginal and transdermal hormone delivery methods 4. Intrauterine device (with or without hormone elution)
* Clinically acceptable methods of birth control

  1. Male or female condom with or without spermicide
  2. Norethindrone-based progestin-only oral contraceptives
  3. Cap, diaphragm, sponge with spermicide.

  23. Participation in any clinical trial within 30 days prior to the screening visit.

  24. Change in residence between geographical regions since the last birch pollen season or anticipated relocation away from the geographical region during the pre-determined birch pollen seasons for more than 2 weeks.

  25. Patients who are non-compliant and/or uncooperative, in the Investigator's opinion.

  26. Possible dependency of the patient or patients' parents/authorised legal representative(s) on Sponsor or Investigators/sub-Investigators or trial personnel.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 553 (Actual)
Dates: Start 2023-09-20 (Actual); Primary Completion 2025-08-06 (Actual); Study Completion 2025-08-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint will be the average ARC Total Combined Score (TCS) (TCS0-38) over the entire Birch Pollen Season (BPS) 2. | Following visits after starting the study: at 16 months, 18 months
  The Average Adjusted Symptom Score (AadSS(0-18)) a score based on the daily Rhino-conjunctivitis Total Symptom Scores (RTSS) and adjusted for the daily rescue medication (RM) usage, while on treatment during the BPS2.

SECONDARY OUTCOMES:
The average CSMS (CSMS0-6) | Following visits after starting the study: at 16 months, 18 months
  The average CSMS0-6 is an average of the non-missing daily CSMS0-6, with CSMS0-6 defined as CSMS0-6= DSS0-3 +DMS0-3.
  * The DSS0-3 is calculated as the average of the scores for each individual ARC symptom (runny nose, blocked nose, sneezing, itchy nose, itchy eyes, watery eyes).
  * The DMS0-3 is based on rescue medication intake and ranges from 0 to 3 with:
    * 0=No rescue medication taken,
    * 1=Patient took antihistamine (eye drops and/or oral form),
    * 2=Patient took nasal corticosteroid,
    * 3=Patient took oral corticosteroid as a concomitant treatment to manage asthma exacerbation, if the case arises.
The average ARC DSS (DSS0-18) | Following visits after starting the study: at 16 months, 18 months
  The average DSS0-18 is calculated as the average of the daily (non-missing) DSS0-18
The average ARC DMS (DMS0-20) | Following visits after starting the study: at 16 months, 18 months
  The average DMS0-20 calculated as the average of the daily (non-missing) DMS0-20
The overall RQLQ(S) score | Following visits after starting the study: at 16 months, 18 months
  The overall RQLQ(S) score calculated as the mean of responses.
The overall PRQLQ score | Following visits after starting the study: at 16 months, 18 months
  The overall PRQLQ score calculated as the mean of responses.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Pfarr, MD, Principal Investigator — Department of Otorhinolaryngology, Head and Neck Surgery, University Hospital Marburg
Locations (61):
- Austria (3):
  - VIENNA GENERAL HOSPITAL / Medical University of Vienna, Vienna
  - Allergie Ambulatorium, Vienna
  - Allergie Zentrum Wien West, Vienna
- Bulgaria (4):
  - UMHAT Sveti Georgi EAD, Plovdiv
  - Acibadem City Clinic Tokuda Hospital, Sofia
  - DCC NeoClinic, Sofia
  - MC Hera, Sofia
- Finland (2):
  - Terveystalo Jyvaskyla, Jyväskylä
  - Terveystalo Hospital, Tampere
- Alyatec, Strasbourg, France
- Germany (10):
  - Universitaesklinikum Augsburg, Augsburg
  - FA f. Hals-Nasen-Ohrenheilkunde Berlin, Berlin
  - HNO Praxis Dreieich, Dreieich
  - Praxisklinik am Altmarkt / Studienzentrum Dresden, Dresden
  - Yarin Yury, Dr.med., Dresden
  - HNO-Praxisgemeinschaft Dr. med. Frank Bohm/ Marcus Hochhaus, Hannoversch Münden
  - Universitätsklinikum Marburg, Marburg
  - Hno-Praxis Dr. Med. Sonja Runge, Neuenhagen
  - HNO research GmbH / HNO im Norden MVZ, Rendsburg
  - Zentrum fuer Rhinologie und Allergologie - Wiesbaden, Wiesbaden
- Hungary (4):
  - DRC Gyogyszervizsgalo Kozpont Kft., Balatonfüred
  - Clinexpert Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont Infektologiai Klinika, Debrecen
  - Somogy Megyei KAposi Mor Oktato Korhaz, Kaposvár
- Latvia (5):
  - Association of Balvu and Gulbene Hospitals, Balvi
  - Private practice of pneimology and alergology, Rēzekne
  - The Centre of Investigation and Treatment of Allergyc Diseases, Riga
  - Children CUH, Riga
  - LOR Clinic, Riga
- Lithuania (7):
  - CD-8 Clinic Kaunas, Kaunas
  - Vsj Respublikine Siauliu Ligonine, Šiauliai
  - Mama, As Sergu, Vilnius
  - Inovatyvios Alergologijos Centras, Vilnius
  - JSC, Center for Diagnosis and Treatment of Allergic Diseases, Vilnius
  - SEIMOS GYDYTOJAS Vaiku ligonine Vsl Vilniaus universiteto ligonines Santariskiu kliniku filialas, Vilnius
  - Ausveja Uab, Vilnius
- Poland (15):
  - Allergy Clinic Homeo Medicus, Bialystok
  - Clinical Trials Medical Practice, Bialystok
  - Gabinet Prywatna Praktyka Lekarska, Bialystok
  - Clinica Vitae, Gdansk
  - Indywidualna Specjalistyczna Praktyka Lekarska Elzbieta Matusz, Gryfice
  - Vita Longa Sp. z o.o., Katowice
  - Centrum Medyczne PLEJADY, Krakow
  - ETG Lodz, Lodz
  - Alergotest 5C. Specjalistyczne Centrum Medyczne, Lublin
  - Makowskie Centrum Medyczne Hamernia, Maków
  - Centrum Alergologii w Poznaniu, Poznan
  - SNZOZ AlergologaPlus, Poznan
  - Irmed Centrum Alergologii, Warsaw
  - All-Med Specjalistyczna Opieka Medyczna. Medyczny Instytut Badawczy, Wroclaw
  - PROXIMUM, Wroclaw
- Spitalul Clinic de Urgenta pentru Copii Grigore Alexandrescu, Bucharest, Romania
- Slovakia (6):
  - Alergoimuno centrum s.r.o., Kežmarok
  - Alersa s.r.o., Košice
  - Pneumoimunoalergologicka ambulancia Klinika deti a dorastu Martinska fakultna nemocnica, Martin
  - ProbarE Lund, Prešov
  - Zoll - Med - s.r.o, Rimavská Sobota
  - Ambulancia klinickej imunologie a alergologie, Šurany
- Sweden (3):
  - Delta Health Care SRL, Linköping
  - Delta Health Care SRL, Lund
  - Delta Health Care SRL, Stockholm